CLINICAL TRIAL: NCT04535128
Title: COVID-19 Registry to Assess Frequency, Risk Factors, Management, and Outcomes of Arterial and Venous Thromboembolic Complications (CORONA-VTE NET)
Brief Title: COVID-19 Registry to Assess Frequency, Risk Factors, Management, and Outcomes of Arterial and Venous Thromboembolic Complications
Acronym: CORONA-VTE NET
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry); University of Colorado, Denver (Other); Anne Arundel Medical Center (Individual); Beth Israel Deaconess Medical Center (Other); Jefferson Medical College of Thomas Jefferson University (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Other Study IDs: 2020P000848
Record Dates: First submitted 2020-08-29; First posted 2020-09-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Covid19; Thrombosis Embolism; DVT; Pulmonary Embolism; Myocardial Infarction; Stroke
Keywords: COVID-19; Thromboembolism
MeSH Terms: conditions — COVID-19; Embolism and Thrombosis; Pulmonary Embolism; Myocardial Infarction; Stroke; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Positive: Patients with positive COVID-19 PCR
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Novel coronavirus 2019 (COVID-19) has emerged as a major international public health concern. While much of the morbidity and mortality associated with COVID-19 has been attributed to acute respiratory distress syndrome (ARDS) or end-organ failure, emerging data suggest that disorders of coagulation, in particular hypercoagulability and venous thromboembolism (VTE), may represent an additional major, and possibly preventable, complication (Wu C, et al. JAMA Intern Med. 2020 Mar 13. [Epub ahead of print] and Tang N, et al. Thromb. Haemost. 2020 Feb 19. [EPub Ahead of Print]). Abnormal coagulation testing results, especially markedly elevated D-dimer and FDP, have been associated with a poor prognosis in COVID-19 infection. We propose the following Electronic Health Record (EHR)-guided 10000-patient, retrospective observational cohort study to assess VTE incidence, risk factors, prevention and management patterns, and thrombotic outcomes in patients with COVID-19 infection. In order to gain the valuable perspective of other regional and national centers providing care for large populations of COVID-19, we have started a collaborative network with 5 additional sites which will provide us with de-identified data from 1000 patients each. These 5000 patients in addition to the 5000-patient cohort we are enrolling within the Mass General Brigham Network will comprise this study population.

DETAILED DESCRIPTION:
Aim #1: To determine the 30-day and 90-day frequencies of adjudicated, symptomatic arterial and venous thromboembolic events in patients with COVID-19 infection. Symptomatic VTE is defined as symptomatic DVT or PE, confirmed by imaging, within 30 days of randomization. Arterial thromboembolism will be comprised of myocardial infarction, stroke or systemic embolism, acute limb ischemia.

Aim #2: To determine VTE-related risk factors, prevention and management patterns, and 30-day and 90-day all-cause mortality, bleeding, and thrombotic outcomes in patients with COVID-19 infection. 30- and 90-day bleeding outcomes will include ISTH-major and clinically-relevant nonmajor bleeding. Thrombotic outcomes will include symptomatic VTE, myocardial infarction, stroke or systemic embolism, acute limb ischemia, and cardiovascular death.

Aim #3: To determine through multivariate logistic regression modeling, independent risk factors for VTE in patients with COVID-19 infection that could be used to identify those who may benefit from thromboprophylaxis during hospitalization and after discharge.

Study Design: 10000 patient U.S.-based EHR-guided, retrospective observational cohort analysis. Data will abstracted through the EHR. Because this is a computer-generated observational retrospective registry, informed consent will not be practical. Accordingly, we will ask our Institutional Review Board to waive the requirement for informed consent. Participating sites (University of Colorado, Jefferson Health, BIDMC, Anne Arundel Medical Center, and another site to be named) will obtain IRB approval at their own institutions.

Study Population: Patients are eligible if they are ≥18 years of age and meet the following criteria:

1. Positive COVID-19 PCR AND
2. Inpatient OR outpatient management of COVID-19 infection

Patient Enrollment: We will create a search engine query through the EHR to identify patients with an objective COVID-19 diagnosis who are hospitalized or being treated as outpatients. This will be executed retrospectively for patients already objectively-diagnosed at participating clinical sites.

Primary Outcome: 30-day and 90-day frequency of objectively confirmed, adjudicated arterial thromboembolism or VTE, including deep venous thrombosis (DVT) and pulmonary embolism (PE).

Secondary Outcome: 30-day and 90-day frequency of adjudicated all-cause death, bleeding, and thromboembolic outcomes.

Additional Variables of Interest: Additional measured variables will include VTE-related risk factors, prevention and management patterns, and cause of death. We will review the notes and diagnostic testing sections of the Electronic Health Record to complete an electronic case report form for each subject.

Follow-Up: Follow-up will consist of Electronic Health Record review at 30 days and 90 days from study entry.

ELIGIBILITY:
1. Positive COVID-19 PCR AND
2. Inpatient OR outpatient management of COVID-19 infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with documented COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of arterial or venous thromboembolism over 30 days | 30 days
  Frequency (%) of arterial or venous thromboembolism
Frequency of arterial or venous thromboembolism over 90 days | 90 days
  Frequency (%) of arterial or venous thromboembolism

SECONDARY OUTCOMES:
Frequency of all-cause death, bleeding, and thromboembolic outcomes at 30 days | 30 days
  Frequency (%) of all-cause death, bleeding, and thromboembolic outcomes
Frequency of all-cause death, bleeding, and thromboembolic outcomes at 90 days | 90 days
  Frequency (%) of all-cause death, bleeding, and thromboembolic outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, MD, MS, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No